CLINICAL TRIAL: NCT02185768
Title: Chemoembolisation of Hepatocellular Carcinomas Not Subject to Interventive Care by Idarubicin-loaded Beads - IDASPHERE II
Acronym: IDASPHERE II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1307
Record Dates: First submitted 2014-07-03; First posted 2014-07-10 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Liver Cancer
Keywords: Liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC-BEADS + Idarubicin (Experimental): Chemoembolization with DC BEAD loaded with idarubicin
  Interventions: Drug: idarubicin; Device: Dc- Beads 300-500µm

INTERVENTIONS:
Drug: idarubicin
Device: Dc- Beads 300-500µm

SUMMARY:
The most frequently used products in CHE are doxorubicin (36%), cisplatin (31%), and epirubicin (12%). But until recently, there were no obvious reasons to use one product over another. In fact, systemic chemotherapy is considered ineffective in HCC [hepatocellular carcinoma], which does not allow any argument in favour of the product. Moreover, 2 randomised trials comparing the molecules (doxorubicin vs. epirubicin) proved to be negative in terms of survival.

Cytotoxicity of different anticancer agents on HCC cell lines have been compared in order to select the best candidate for CHE. Eleven chemotherapy molecules have been tested, including those more frequently used in CHE. Among them, idarubicin (an anthracycline) proved to be the most effective in vitro by far. The superiority of idarubicin (as opposed to doxorubicin) was noted especially on the SNU-449 line, which is known for its resistance to several chemotherapy agents. The best cytotoxicity of idarubicin can be explained by 2 mechanisms: 1) idarubicin has a better intracellular penetration than the other anthracyclines. This is probably due to its more considerable lipophily, facilitating thus its passage through the membrane made up of a double lipid layer, 2) idarubicin is resistant to the multidrug resistance system (MDR). The MDR mechanism, which is often noted in HCC, consists of membrane pumps transporting the molecule outside the cell. These two particularities could explain a more significant accumulation of idarubicin in the HCC cells, and thus better efficacy. It is interesting to note that orally administered idarubicin (5 mg/day for 21 days) has proved to be less toxic and is effective in HCC. Currently, idarubicin is used to treat leukaemia. Its toxicity profile (especially, haematological and cardiac) is known.

On these grounds, A pilot study has been conducted in order to assess the tolerance and efficacy of lipiodol-based CHE using a 10 mg dose of idarubicin in 21 patients with unresectable HCC. These preliminary data reveal that CHE with idarubicin is effective and less toxic.

Idarubicin can be loaded in microbeads. A phase I study (IDASPHERE) has been conducted on DC Beads® microbeads (300-500µm) loaded with idarubicin (dose increased from 5 to 25 mg). The DLT [dose-limiting toxicity] and MTD [maximum tolerated dose] have been determined in 21 patients using a CRM. The MTD of idarubicin was assessed at 10 mg. In our study, the idarubicin-loaded beads did not give rise to any specific toxicity-related problem. The 10 mg dose is compatible with the known toxicity profile of idarubicin: cumulative cardiotoxicity of doxorubicin is noted from 550 mg/m², whereas that of idarubicin is noted from 93 mg/m². There is thus a 5.9:1 ratio between their cumulative toxicities. The most frequently used dose (and also the weakest one) for the doxorubicin-based CHE is 50 mg. The equivalent of the idarubicin dose would thus be: 50 mg (doxorubicin) / 5.9 (doxorubicin/idarubicin ratio) = approx. 10 mg of idarubicin.

It has been already demonstrated that hepatic extraction of idarubicin is better than those of doxorubicin and daunorubicin in an animal sarcoma model. In this study, AUC 0-48h and AUC 0-72h were 1.35 times higher with idarubicin, proving that its intra-hepatic penetration was 35% higher.

The randomised phase II PRECISION V study compared conventional CHE (cCHE) with CHE by doxorubicin beads (DC Bead®) in patients with HCC. It is currently the largest randomised trial on CHE published. The PRECISION V data can be thus used to compare the other studies in terms of efficacy and tolerance.

To continue our preliminary study and the phase I IDASPHERE study, investigators wish to assess thus the efficacy and confirm the tolerance of idarubicin-loaded beads for the CHE of HCC according to a protocol similar to PRECISION V, as part of a single-arm phase II study.

DETAILED DESCRIPTION:
By using a 2-step Fleming plan (Fleming, 1982) with a unilateral alpha risk of 5% and 90% potency, it is necessary to include 86 assessable patients.

On the 1st step: 43 patients will be included (+/- 2 patients, if non-assessable patient(s)

* If 10 patients or less present an objective response, the trial will be discontinued on grounds of futility (H1 rejected)
* If 18 patients or less present an objective response, the trial will be discontinued on grounds of efficacy (H0 rejected)

If not, we proceed with the 2nd step including 43 additional patients. If 29 patients or more present an objective response, the treatment will be considered as effective (H0 rejected)

Considering a 5% ratio of visual loss or non-assessable patients, 91 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* - Histologically diagnosed HCC or HCC diagnosed according to the EASL criteria
* Measurable targets according to the mRECIST v1.1 criterion
* Preserved liver function (in case of Child-Pugh A or B7 cirrhosis)
* Tumour not subject to interventive care (liver transplant, surgical resection or percutaneous destruction)
* BCLC A/B without portal or extra-hepatic invasion
* No prior treatment by chemotherapy, radiotherapy or transarterial embolisation (with or without chemotherapy)
* Age ≥ 18 years
* WHO 0 or 1
* Laboratory test: platelets ≥ 50,000 mm3, N ≥ 1,000/mm3, creatininaemia ≤ 150 µmol/L, PT ≥ 50%
* No heart failure (isotope or ultrasound VEF > 50%)

Exclusion Criteria:

* - Advanced tumour (vascular or extra-hepatic invasion including brain metastasis or diffuse HCC with liver invasion > 50%)
* History of other type of cancer except cancer known to be in remission for more than 5 years (in this case, HCC histological proof is required), or basal-cell carcinoma or in situ cervix uteri cancer properly treated with curative treatment
* Advanced liver disease (Child B8, B9 and C, bilirubinaemia > 3 mg/dL, SGOT and SGPT > 5 x ULN or 250 U/L)
* Previous treatment by idarubicin and/or doxorubicin
* Idarubicin contraindications (cardiopathy with myocardial failure, serious kidney or liver failure, yellow fever vaccine)
* Concurrent disease or uncontrolled severe clinical condition
* Uncontrolled severe infection
* Patient requiring long-term anticoagulant treatment
* Thrombosis of the portal vein or a 3-segment region or more
* Hepatofugal portal venous flow
* Presence of serious atheromatosis
* Presence of collateral vascular ways potentially affecting the normal regions during embolisation
* Presence of arthritis of the hepatic artery branches to be treated
* Presence of arterioportal or arterial subhepatic fistula that cannot be embolised by coils
* Pregnancy or breastfeeding
* Absence of effective contraception (for men and women of childbearing age)
* Patient who cannot be regularly monitored on account of psychological, social, family- or geography-related reasons
* Concomitant participation of a patient in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris GUIU, PhD, Principal Investigator — Fédération Francophone de Cancérologie Digestive
Locations (7):
- France (7):
  - CHU Amiens, Amiens
  - CHU d'ANGERS, Angers
  - CHU - Hôpital François Mitterand, Dijon
  - Hôpital La Croix Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - CHU St Eloi, Montpellier
  - Hôpital de l'Archet II, Nice

REFERENCES:
- [Result] Guiu B, Chevallier P, Assenat E, Barbier E, Merle P, Bouvier A, Dumortier J, Nguyen-Khac E, Gugenheim J, Rode A, Oberti F, Valette PJ, Yzet T, Chevallier O, Barbare JC, Latournerie M, Boulin M. Idarubicin-loaded Beads for Chemoembolization of Hepatocellular Carcinoma: The IDASPHERE II Single-Arm Phase II Trial. Radiology. 2019 Jun;291(3):801-808. doi: 10.1148/radiol.2019182399. Epub 2019 Apr 30. PMID 31038408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-six patients were included by 7 centers between January 2015 and June 2016.
Groups:
- DC-BEADS + Idarubicin: Two vials of 100-300 μm of drug-eluting beads (DC Bead) were loaded with 10 mg of idarubicin in aseptic conditions at the hospital pharmacies prior to TACE. Rapidly, 10 mg of idarubicin were reconstituted with 5 mL of sterile water for injection. As much saline as possible was removed from the two vials to add 5 mg (ie, 2.5 mL) of idarubicin. After a loading time of 60 minutes, the solution containing idarubicin-loaded beads was transferred to a 30-mL syringe. Just before injection, the interventional radiologists added 5 mL per milliliter of beads of a nonionic contrast medium to the syringe containing idarubicin-eluting beads. It was recommended to use 2.4-F to 2.8-F microcatheters for the catherization of tumor feeders, to perform cone-beam CT as soon as deemed necessary, and to inject the beads slowly (ideally 1 mL/min) through a 1-mL syringe until either complete delivery of the beads or reduced flow of the feeding artery with the conventional method of two to five heartbeats to clear the contrast column from the microcatheter tip.
Period: Overall Study
Arm/Group | DC-BEADS + Idarubicin
Started | 46
Completed | 44 (corresponding to the mITT population)
Not Completed | 2
Not completed — Patients were not treated | 2

BASELINE CHARACTERISTICS:
Population: Baseline data are done on the ITT population meaning all the patients included in the study
Groups:
- DC-BEADS + Idarubicin: Chemoembolization with DC BEAD loaded with idarubicin
  idarubicin
  Dc- Beads 300-500µm
Arm/Group | DC-BEADS + Idarubicin
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.25 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response or Partial Response (Objective Response), as Assessed According Central Review
Description: The main judgement criterion is the rate of patients in objective response (complete or partial response) at 6 months according to the mRECIST criteria and based on the central review. Response Evaluation Criteria In Solid Tumors Criteria (mRECIST v1.0) for target lesions was assessed by MRI Complete Response (CR) was defined as : Disappearance of all target lesions and Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response was defind as the number of patients with a CR or a PR.
Time Frame: up to 6 months
Population: The modified intention-to-treat (mITT) population was defined as all evaluable patients included in the study regardless of eligibility criteria. A patient was considered evaluable if the patient had at least one chemoembolization and one post-treatment evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | DC-BEADS + Idarubicin
Number analyzed (Participants) | 44
Participants
  Objective response | 22
  No objective response | 22

2. Secondary Outcome: Number of Participants With Complete Response or Partial Response (Objective Response), as Assessed by the Investigator
Description: The rate of patients in objective response (complete or partial response) at 6 months according to the mRECIST criteria, and assessed according to the investigator. Response Evaluation Criteria In Solid Tumors Criteria (mRECIST v1.0) for target lesions wasassessed by MRI Complete Response (CR) was defined as : Disappearance of all target lesions and Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response was defind as the number of patients with a CR or a PR.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DC-BEADS + Idarubicin
Number analyzed (Participants) | 44
Participants
  Complete response | 12
  Partial response | 8
  Stability | 0
  Progression | 23
  Non evaluable | 1

3. Secondary Outcome: Best Response According to mRECIST v1.0 in MRI
Description: The best response according to the mRECIST criteria. Response Evaluation Criteria In Solid Tumors Criteria (mRECIST v1.0) for target lesions was assessed regarding all MRI done for patient during its treatment period.
Time Frame: up to 6 months after last chemoembolisation
Measure: Count of Participants; unit: Participants
Arm/Group | DC-BEADS + Idarubicin
Number analyzed (Participants) | 44
Participants
  Complete response | 17
  Partial response | 13
  Stability | 8
  Progression | 5
  Non evaluable | 1

4. Secondary Outcome: Progression-Free Survival
Description: It was defined by the time interval between the inclusion date and the date of the 1st progression according to the mRECIST criteria (assessed in central review) or death (regardless of the cause).
  Alive patients without progression were censored at date of the last news.
Time Frame: up to 2 years
Population: Analysis was done on the ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DC-BEADS + Idarubicin
Number analyzed (Participants) | 46
months | 6.57 [5.85 to 11.99]

5. Secondary Outcome: Overall Survival
Description: It was defined by the time interval between the inclusion date and date of death (regardless of the cause) or date of the last news for alive patients.
Time Frame: up to 3 years
Population: Analysis was done on the ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DC-BEADS + Idarubicin
Number analyzed (Participants) | 46
months | 18.55 [11.73 to 29.08]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment. The mean treatment duration was 6 months. After the definitive stop of the protocol, patients were only followed-up for the overall survival up to 3 years
Arm/Group | DC-BEADS + Idarubicin
All-Cause Mortality (participants affected / at risk) | 32/46
Serious Adverse Events (participants affected / at risk) | 15/46
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DC-BEADS + Idarubicin (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Ascite (Gastrointestinal disorders) | 1 (1)
Upper GI haemorrhage (Gastrointestinal disorders) | 1
Varices Oesophageal (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Biloma (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Bacteraemia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Post-embolisation syndrome (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anxiety (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Malignant hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DC-BEADS + Idarubicin (N=44)
Cephalgia (Nervous system disorders) | 3
Stomach pain (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Anemias (Blood and lymphatic system disorders) | 16
Hypertension (Vascular disorders) | 4
Pain (General disorders) | 15
Alanine aminotransferase increased (Investigations) | 31
Aspartate aminotransferase increased (Investigations) | 33
Total Bilirubin increased (Investigations) | 28
Creatinine increased (Investigations) | 5
Gammaglutamyltransferase increased (Investigations) | 27
White blood cell count decreased (Investigations) | 4
Lipase increased (Investigations) | 4
Neutropenia (Investigations) | 4
Lymphocytes decreased (Investigations) | 12
Phosphatases alcalines increased (Investigations) | 16
Platelets decreased (Investigations) | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 23
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 21
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypokaliemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Asthenia (General disorders) | 8
Fever (General disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT02185768/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT02185768/SAP_001.pdf